CLINICAL TRIAL: NCT05123612
Title: Effects of Fermented & Fiber-rich Foods on Maternal & Offspring Microbiome Study
Brief Title: Maternal & Offspring Microbiome Study
Acronym: MOMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Rehnborg Farquhar Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 61806
Record Dates: First submitted 2021-10-27; First posted 2021-11-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related; Microbiome; Immune Function; Inflammation
Keywords: Pregnancy; Microbiome; Immune function; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Dietary Fiber; Fermented Foods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fiber (Experimental): Participants will be asked to increase their usual dietary fiber intake by 20 grams/day.
  Interventions: Behavioral: Fiber
- Fermented Foods (Experimental): Participants will be asked to consume 6 servings of fermented foods per day.
  Interventions: Behavioral: Fermented Foods
- Fiber + Fermented Foods (Experimental): Participants will be asked to increase their usual dietary fiber intake by 20 grams/day and to consume 6 servings of fermented foods per day.
  Interventions: Behavioral: Fiber; Behavioral: Fermented Foods
- Comparator (No Intervention): Participants will receive usual care for pregnancy and postpartum.

INTERVENTIONS:
Behavioral: Fiber — Additional 20 grams of fiber/day.
  Arms: Fiber; Fiber + Fermented Foods
Behavioral: Fermented Foods — 6 servings of fermented foods/day
  Arms: Fermented Foods; Fiber + Fermented Foods

SUMMARY:
The purpose of the study is to learn how different dietary interventions affect microbiota diversity in pregnant women and the transmission of microbiota to their infants during pregnancy, birth, and postpartum.

DETAILED DESCRIPTION:
This research study aims to understand the relationship of dietary fiber, fermented foods, and the microbiome, specifically during pregnancy and postpartum. The investigators know that the composition of the microbiome can have an important effect on overall health, and a greater variety will confer more health benefits. Research suggests that maternal microbiota play an important role in the development of their offspring's microbiota during pregnancy, childbirth, and breastfeeding. The purpose of this study is to assess how diet impacts maternal microbiome during pregnancy and their infant's microbiome up to about two years postpartum.

Potential pregnant participants will be recruited during their first trimester up to 22 weeks. After completion of the baseline visit and sample collection, they will be randomized to start a diet high in fiber, high in fermented foods, high in both fiber and fermented foods, or a usual care group. Participants will be asked to provide blood, stool, vaginal swab, and breast milk samples periodically throughout the study. Cord blood will be collected after childbirth, and infant blood from a heel stick will be collected twice. They will also be asked to fill out online questionnaires and perform dietary recalls with study diet assessors.

After completing the study, participants will be invited to continue to participate in an extension of the study for approximately three and a half additional years. The purpose of this extension is to continue to assess how diet impacts the mother's microbiome postpartum and the child's microbiome up to about 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Singleton pregnancies
* Recruit during the first trimester and up to 22 weeks of pregnancy.
* Healthy subjects willing and able to provide blood, stool, vaginal swab, and breast milk samples.
* Must be able to provide signed and dated informed consent.

Exclusion Criteria:

* Pre-pregnancy BMI greater than 40
* Blood pressure SBP: > 160 mmHg -OR- DBP: > 90 mmHg
* Kidney disease
* Liver disease
* Anemia
* Symptomatic gallstones
* History of bariatric surgery
* Acute disease at time of enrollment (i.e. flu or gastroenteritis). May delay sampling until subject recovers.
* Chronic, clinically significant, unstable (unresolved, requiring on-going changes to medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history
* History of active uncontrolled gastrointestinal disorders or diseases including:
* Inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis;
* Irritable bowel syndrome (IBS) (moderate-severe);
* Persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated)
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection.
* Surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* Confirmed or suspected autoimmune disease

Medications:

* Weight loss medications
* Regular high dose aspirin
* Regular use of prescription opiate pain medication

If taken in the past 2 months:

* Systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular or oral)
* Corticosteroids (intravenous, intramuscular, oral, nasal or inhaled)
* Cytokines
* Methotrexate or immunosuppressive cytotoxic agents

Diet & Lifestyle:

* Recent history of chronic excessive alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day; or > 14 drinks/week.
* Regular/frequent use of smoking or chewing tobacco, e-cigarettes, cigars or other nicotine-containing products

Maternal chronic medical conditions:

* Pre-gestational diabetes (T1 or T2)
* History of gestational diabetes
* On medication that is an immune modulators or chronic steroid use
* Hyperemesis gravidarum

Pregnancy history:

* Preterm birth
* Recurrent pregnancy loss

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 135 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2029-09-09 (Estimated); Study Completion 2029-09-09 (Estimated)

PRIMARY OUTCOMES:
Difference in total number of species detected in stool as a measure of infant microbiota diversity. | 1 month postpartum
  Difference in total number of species (ASVs - Amplicon Sequence Variants) detected in stool between the fiber, fermented, fiber + fermented and comparator arms at 1 month postpartum.

SECONDARY OUTCOMES:
Change in the total number of species detected in stool as a measure of maternal microbiota diversity. | Baseline and 36 weeks of pregnancy
  Change in differences in total number of species (ASVs- Amplicon Sequence Variants) detected in stool from baseline to 36 weeks of pregnancy between fiber, fermented, fiber + fermented, and comparator arms.
Change in the maternal inflammatory marker profile | Baseline and 36 weeks of pregnancy
  Change in the differences in inflammatory markers (β-NGF, LIF-R, IL-12B, IL10, CASP-8, LAP TGF-β-1, CD6, CD5, MCP-2, IL6, CCL20, IL18, VEGFA, MMP-10, MCP-4, CCL4, CXCL10, CCL19, FGF-21) detected in blood samples from baseline to 36 weeks of pregnancy between fiber, fermented, fiber + fermented, and comparator arms.
Characterize the infant inflammatory marker profile | 6 months postpartum
  Difference in amount of inflammatory markers (β-NGF, LIF-R, IL-12B, IL10, CASP-8, LAP TGF-β-1, CD6, CD5, MCP-2, IL6, CCL20, IL18, VEGFA, MMP-10, MCP-4, CCL4, CXCL10, CCL19, FGF-21) detected in heel stick blood between fiber, fermented, fiber + fermented, and comparator arms at 6 months postpartum.
Characterize the infant allergy marker profile | 6 months postpartum
  Difference in amount of allergy markers (skin prick testing) detected in heel stick blood between fiber, fermented, fiber + fermented, and comparator arms at 6 months postpartum.
Infant Growth | 18 months postpartum
  Difference in weight-for-length growth chart percentiles between fiber, fermented, fiber + fermented, and comparator arms at 18 months postpartum.
Maternal Weight | 36 weeks of pregnancy
  Differences in the number of participants who gained weight within the pregnancy weight gain recommendations between fiber, fermented, fiber + fermented, and comparator arms measured at 36 weeks.
Maternal systolic blood pressure | Baseline and 36 weeks of pregnancy
  Change from baseline in systolic blood pressure at 36 weeks of pregnancy.
Maternal diastolic blood pressure | Baseline and 36 weeks of pregnancy
  Change from baseline in diastolic blood pressure at 36 weeks of pregnancy.
Maternal LDL-cholesterol | Baseline and 36 weeks of pregnancy
  Change from baseline in LDL cholesterol at 36 weeks of pregnancy.
Maternal HDL-cholesterol | Baseline and 36 weeks of pregnancy
  Change from baseline in HDL cholesterol at 36 weeks of pregnancy.
Maternal triglycerides | Baseline and 36 weeks of pregnancy
  Change from baseline in triglycerides at 36 weeks of pregnancy.
Maternal glucose | Baseline and 36 weeks of pregnancy
  Change from baseline in glucose at 36 weeks of pregnancy.
Maternal fasting insulin | Baseline and 36 weeks of pregnancy
  Change from baseline in fasting insulin at 36 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Garnder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ward CP, Perelman D, Durand LR, Robinson JL, Cunanan KM, Sudakaran S, Sabetan R, Madrigal-Moeller MJ, Dant C, Sonnenburg ED, Sonnenburg JL, Gardner CD. Effects of fermented and fiber-rich foods on maternal & offspring microbiome study (FeFiFo-MOMS) - Study design and methods. Contemp Clin Trials. 2025 Mar;150:107834. doi: 10.1016/j.cct.2025.107834. Epub 2025 Feb 1. PMID 39900290
- See also: Study description — https://med.stanford.edu/nutrition/research/current-studies/fefifo-moms.html